CLINICAL TRIAL: NCT02104440
Title: Clinical Trial In The Treatment Of Allogeneic Post-Transplant Cytopenias With Sequential Infusion Of Allogeneic Mesenchymal Cells Expanded In Vitro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: University of Navarrra Hospital (Clinica Universitaria) (Other); Haematology Service,University Hospital of Salamanca, MªConsuelo del Cañizo Fernández-Roldán (Other); Hospitales Universitarios Virgen del Rocío (Other); Spanish National Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/CIT; 2013-000534-35 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-04-04 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Cytopenia
Keywords: Cytopenia
MeSH Terms: conditions — Cytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with cytopenia after allo-HSCT (Experimental): Patients with cytopenia after allo-HSCT
  Interventions: Biological: Sequential infusion of allogeneic mesenchymal stem cells expanded "in vitro"

INTERVENTIONS:
Biological: Sequential infusion of allogeneic mesenchymal stem cells expanded "in vitro"

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the sequential infusion of allogeneic mesenchymal stem cells (MSC), expanded "in vitro" with platelet lysate without addition of animal products in the treatment of patients undergoing allo-HSCT who developed one or more cytopenias.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies who have been subjected to allo-HSCT and that are diagnosed with one or more peripheral cytopenias with complete chimerism in bone marrow (determined by molecular-STR-studies). They may include:

  1. Patients who have received as a source of cells MO or SP
  2. Patients who have received cells from a related donor or unrelated HLA-matched
  3. Patients transplanted with myeloablative or non-myeloablative conditioning
* Adequate cardiac function assessed from a clinical point of view by the researcher, with no history of ischemic heart disease (angina or myocardial infarction) in the previous 6 months.
* Adequate pulmonary function assessed clinically without evidence of severe obstructive or restrictive lung disease.
* Patients between 18 and 70 years
* Signed informed consent

Exclusion Criteria:

* Patients whose haemopathy has not been controlled by the transplantation or is in progress at the time of treatment.
* Patients who do not have complete chimerism in bone marrow (performed within 28 days prior to baseline by molecular study -STR-).
* Patients with thrombotic microangiopathy.
* Patients with post-transplant cytopenias with toxic origin in relation to antiviral treatment (eg ganciclovir, valganciclovir) without concomitant graft against host disease.
* Patients with bacterial, viral or fungal infection that is not being controlled with proper treatment.
* Patients with a history of ischemic heart disease (angina or myocardial infarction) in the previous 6 months, and those considered by the investigator does not have adequate cardiac function, evaluated from a clinical point of view.
* Patients with poor lung function, evaluated clinically, according to the researcher.
* Patients who, in the opinion of the investigator, are not on a good position to tolerate treatment.
* Patients who do not have the required donor.
* Women pregnant or at risk of pregnancy by contraceptive measures inadequate.
* Patients <18 or > 70 years.
* Patients who did not sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Adverse effects at the time of infusion and infections after infusion of MSC | During the period of infusion of the cells into the patient (an average of one hour)
  All the adverse effects that may arise and possible toxicities (WHO grade) after infusion of the cells were collected.

SECONDARY OUTCOMES:
Mesenchymal cell efficiency in recovering cytopenia | Monitoring will be from the last infusion of MSCs to the patient until 90 days after the last administration
  The efficiency is measured by the recovery of cytopenia after administration of MSC (depending on the original cytopenia) and may be of two types:
  Complete response:
  * Hb> 10 g / dL
  * Neutrophils> 1500 Million / L
  * Platelets> 100.000 Million / L
  * Maintained at least 7 days
  Partial response:
  * Hb> 8 and <10 g / dL
  * Neutrophils> 1000 and <1500 Million / L
  * Platelets> 50000 and <100.000 Million / L
  * Maintained at least 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Sánchez-Guijo Martín, Ph.D, Principal Investigator — University Clinical Hospital of Salamanca; José Rifón Roca, Ph.D, Principal Investigator — University of Navarrra Hospital (Clinica Universitaria); José A Pérez Simón, Ph.D, Principal Investigator — Hospital Virgen del Rocío
Locations (1):
- University Clinical Hospital of Salamanca, Salamanca, Salamanca/Castilla León, Spain